CLINICAL TRIAL: NCT00987285
Title: Linking Self-Management and Primary Care for Diabetes
Brief Title: Linking Self-Management and Primary Care for Diabetes 2
Acronym: LB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); InterVision (Unknown); Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R01DK035524-21 (NIH); R01DK035524 (NIH)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: RE AIM model; Type 2 Diabetes Mellitus; Interactive voice recognition; Computer Assisted Self Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Computer Assisted Self Management plus Social Support (Experimental): an interactive, automated self-management (ASM) program that uses web and interactive voice recognition (IVR) media combined with enhanced support in the form of group Diabetes Care Management visits and live follow up phone calls from Diabetes Care Managers
  Interventions: Behavioral: CASM +
- Usual care (No Intervention): will receive a health-risk appraisal, interactive CD-ROM program that provides standardized advice on behavior change, but not the hypothesized key intervention processes of goal setting, barriers identification, problem solving, or social environmental support.
- Computer Assisted Self Management (Experimental): An interactive, automated self-management (ASM) program that uses web and interactive voice recognition (IVR) media.
  Interventions: Behavioral: CASM

INTERVENTIONS:
Behavioral: CASM + — Computer Assisted Self Management plus Social Support
  Arms: Computer Assisted Self Management plus Social Support
Behavioral: CASM — Computer Assisted Self Management using and interactive, automated self-management program that uses web and interactive voice recognition (IVR) media
  Arms: Computer Assisted Self Management

SUMMARY:
This project is primarily a behavioral study. We employed a three-arm, patient-randomized practical effectiveness trial to evaluate the impact of two different interactive, multimedia self-management programs, relative to "enhanced" usual care. The two interventions will be (a) the revised program from our present study, based on our social-ecological theory and the 5 As self-management model, plus enhanced support (ASM+ES) that includes practical, but extensive, ongoing support and b) largely Automated Self-Management (ASM). These programs will be compared to a realistic "enhanced usual care" (UC) condition that will provide health risk appraisal feedback, control for computer interactions, and provide standardized advice on behavior change, but not the hypothesized key intervention processes of goal-setting, barriers identification, problem-solving, or social-environmental support. Patients will be randomized to conditions within clinic and will participate for 1 year.

The proposed project will test the effectiveness of a practical, automated-based intervention for primary care patients to facilitate dietary and physical activity practices, and medication-taking. Analyses will focus on primary outcomes of (a) dietary, physical activity, medication-taking outcomes, and (b) the UKPDS risk equation as well as secondary quality-of-life, patient-activation, and patient care outcomes (Specific Aim #2). Using the RE-AIM measures, we will analyze the reach, effectiveness, adoption, implementation, and maintenance of the intervention programs (Specific Aim #3), and also factors related to program implementation, linkage to primary care, and program success with emphasis on cost, cost-effectiveness, and mediators and moderators of outcomes such as social-environment support (Aim #4).

Primary hypotheses:

1. That the Automated Intervention received by Automated self-management (ASM) condition and ASM plus enhanced support conditions (ASM+ES) will be superior to usual care on the primary outcomes.
2. That the ASM+ES condition will be superior to the ASM alone condition on primary outcomes at the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* being 25-75 years of age,
* live independently,
* have a telephone,
* are able to read in either English or Spanish,
* able to access the Internet at least twice per week
* are capable of providing informed consent,
* have been diagnosed with type 2 diabetes for at least 1 year
* are overweight (BMI ≥ 25), and
* have at least one additional UKPDS equation risk factor (i.e., high lipids, hypertension, HbA1c, or smoking)

Exclusion Criteria:

* Exclusion criteria:
* Suffering dementia or active psychosis,
* Being on end-stage dialysis,
* or predicted to live fewer than 2 years
* Being institutionalized.
* Pregnant women - women with gestational diabetes will not be enrolled, because there needs are quite different, but we won't specifically exclude women who are pregnant AND otherwise eligible, since we do acknowledge that it's possible that someone may be unaware that they are pregnant at the time of enrollment, or may become pregnant during the study, and that this will not affect their continued participation.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement in health behaviors (e.g., dietary patterns, physical activity, medication taking) and biologic outcomes (HbA1c, lipid ratio, blood pressure, and smoking status). | Baseline, 4 months and 12 months

SECONDARY OUTCOMES:
Diabetes-specific quality of life (Diabetes Distress Scale), patient activation (PAM scale), and perceived social-environmental support (the Chronic Illness Resources Survey) at 4- and 12-month follow-ups. | 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Glasgow, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente of Colorado, Denver, Colorado, United States

REFERENCES:
- [Background] Glasgow, R.E., Nutting, P.A. (2004) Diabetes. Handbook of Primary Care Psychology. L. Haas (Editor) Oxford University Press, New York, pp 299-319.
- [Background] Glasgow RE, Bull SS, Piette JD, Steiner JF. Interactive behavior change technology. A partial solution to the competing demands of primary care. Am J Prev Med. 2004 Aug;27(2 Suppl):80-7. doi: 10.1016/j.amepre.2004.04.026. PMID 15275676
- [Background] King, D.K., Glasgow, R.E. (2004) Self-management of Type 2 Diabetes: Key Issues, Evidence-Based Recommendations, and Future Directions. In: Best Practices in the Behavioral Management of Chronic Disease, J. Trafton & William Gordon (Eds.). Institute for Disease Management, Los Altos, CA, Vol 2, Chapter 9.
- [Background] Estabrooks PA, Nelson CC, Xu S, King D, Bayliss EA, Gaglio B, Nutting PA, Glasgow RE. The frequency and behavioral outcomes of goal choices in the self-management of diabetes. Diabetes Educ. 2005 May-Jun;31(3):391-400. doi: 10.1177/0145721705276578. PMID 15919639
- [Background] Glasgow RE, Nelson CC, Strycker LA, King DK. Using RE-AIM metrics to evaluate diabetes self-management support interventions. Am J Prev Med. 2006 Jan;30(1):67-73. doi: 10.1016/j.amepre.2005.08.037. PMID 16414426
- [Background] King DK, Estabrooks PA, Strycker LA, Toobert DJ, Bull SS, Glasgow RE. Outcomes of a multifaceted physical activity regimen as part of a diabetes self-management intervention. Ann Behav Med. 2006 Apr;31(2):128-37. doi: 10.1207/s15324796abm3102_4. PMID 16542127
- [Derived] Glasgow RE, Christiansen SM, Kurz D, King DK, Woolley T, Faber AJ, Estabrooks PA, Strycker L, Toobert D, Dickman J. Engagement in a diabetes self-management website: usage patterns and generalizability of program use. J Med Internet Res. 2011 Jan 25;13(1):e9. doi: 10.2196/jmir.1391. PMID 21371992